CLINICAL TRIAL: NCT01486147
Title: Effect of a Visual Nutrient Profiling System on Recall of Nutrition Information
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Nathan Pratt, Mr. Nathan Pratt, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11687 (IRB Protocol #)
Record Dates: First submitted 2011-12-01; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Food labeling; Nutrition; Memory; Diet

ARMS (2):
- Visual (Experimental): Group provided with nutrition information using visual nutrient profiling tool
  Interventions: Behavioral: Visual nutrient profiling tool
- Table (Other): Group provided nutrition information using table format
  Interventions: Behavioral: Nutrient ratings table

INTERVENTIONS:
Behavioral: Visual nutrient profiling tool — Shown color coded fiber and protein 2x2 plot, selected fiber and protein ratings from boxes on the plot.
  Arms: Visual
Behavioral: Nutrient ratings table — Showed nutrition information and had to match to fiber and protein ratings from a table.
  Arms: Table

SUMMARY:
The objective of the study is to validate a visual method of presenting nutritional information by determining if users of the visual method remember food properties better than users given the same information in a non-visual form with texts and tables.

ELIGIBILITY:
Inclusion Criteria:

* Current student at University of Illinois at Urbana-Champaign

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Number of correct responses for fiber and protein ratings of foods | 10 minutes after presentation of nutrition information
  Fiber and protein ratings (5 possible) for 30 foods must be recalled after being presented in a visual or tabular format. Distraction period occurred between presentation of information and recall (maze).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois National Soybean Research Laboratory, Urbana, Illinois, United States